CLINICAL TRIAL: NCT05981690
Title: Therapist Guided, Parent-led, Cognitive Behavioural Therapy (CBT) for Preadolescent Children With Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Kate Harvey, Professor Kate Harvey, University of Reading
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UREC 21/27
Record Dates: First submitted 2023-07-18; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: OCD
Keywords: OCD; CBT; parent

STUDY DESIGN:
Intervention Model Description: Non concurrent multiple baseline design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapist guided, parent-led CBT for preadolescent children with OCD (Experimental): 6 to 8 sessions of therapist guided, parent-led CBT for preadolescent children with OCD
  Interventions: Behavioral: Therapist guided, parent-led CBT for preadolescent children with OCD

INTERVENTIONS:
Behavioral: Therapist guided, parent-led CBT for preadolescent children with OCD — This treatment was adapted from an existing evidence based therapist guided parent-led CBT intervention for preadolescent children with anxiety difficulties. It consists of 6 to 8 treatment individual treatment sessions where parents learn CBT techniques to apply at home with their child

SUMMARY:
This preliminary study aims to examine the outcomes from a therapist guided, parent-led, CBT treatment for preadolescent children (aged 5 to 12 years old) with OCD.

Specifically, this study aims to:

1. Examine outcomes for children who receive the therapist guided, parent-led, CBT treatment for preadolescent children with OCD.
2. Examine parents' experiences and views about the acceptability of the treatment approach.

DETAILED DESCRIPTION:
This study adapted an existing therapist guided, parent-led CBT intervention for children with anxiety difficulties, to ensure suitability for preadolescent children with OCD.

This preliminary study aims to examine the outcomes from a therapist guided, parent-led, CBT treatment for preadolescent children (aged 5 to 12 years old) with OCD.

Specifically, this study aims to:

1. Examine outcomes for children who receive the therapist guided, parent-led, CBT treatment for preadolescent children with OCD.
2. Examine parents' experiences and views about the acceptability of the treatment approach.

ELIGIBILITY:
Inclusion Criteria:

Children

Inclusion criteria:

1. Aged 5 to 12 years old (when parents/carers complete the baseline questionnaires).
2. Diagnosis of OCD (identified from the ADIS-P).
3. UK-resident. Parents

Inclusion criteria:

1. Parent/legal guardian of the child.
2. UK resident.

Exclusion Criteria:

Children

Exclusion criteria:

1. Comorbid condition, which is likely to interfere with treatment delivery, for example:

   1. Established Autism Spectrum Condition (ASC).
   2. Suspected ASC (indicated by exceeding the threshold of 15 on the Social Communication Questionnaire and where a diagnosis of ASC has not been ruled out by a medical professional).
   3. Profound learning difficulty (evidenced by attending a specialist school).
2. Risk and/or safeguarding concerns, which are paramount and would interfere with treatment delivery, for example:

   1. Suicidal intent.
   2. Recurrent or potentially life limiting self-harm.
   3. Significant safeguarding concerns (i.e., if the child has a child protection plan and/or is on the child protection register, and/or the research team consider the child to be suffering, or likely to suffer, significant harm).
3. If children have been prescribed psychotropic medication, the dosage must have been stable for two months.
4. Children who are currently receiving other psychological support/interventions delivered by a mental health professional.

Parents

Exclusion criteria:

1. Significant intellectual impairment that is likely to interfere with treatment delivery.
2. Unable to access or understand written English language materials needed for the intervention.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Children's Yale Brown Obsessive Compulsive Scale (CY-BOCS) | Change from pre-baseline phase, within one-week post-treatment, one-month follow-up
  Diagnostic interview. Higher scores indicate higher severity of OCD

SECONDARY OUTCOMES:
Anxiety Disorder Interview Schedule - Parent Report (ADIS-P) | Change from pre-baseline phase, within one-week post-treatment, one-month follow-up
  Diagnostic interview. Indicates presence/absence of anxiety, OCD, and externalising difficulties. Higher severity scores indicate greater severity of difficulties.
Children's Obsessional Compulsive Inventory - Revised - Parent Report (ChOCI-R-P) | Weekly during baseline and intervention phase; one month follow up
  Symptom measure. Higher scores indicate greater OCD symptoms and impairment.
Family Accommodation Scale - FAS | Weekly during baseline and intervention phase; one month follow up
  Symptom measure. Higher scores indicate greater levels of family accommodation of OCD.
Goal Based Outcomes - GBOs | Weekly during intervention phase; one month follow up
  Families identify up to 3 personalised goals to work towards during the intervention. Goals are rated weekly by the parent form 0 (no goal progress) to 10 (goal achieved)
Session Rating Scale- SRS | Weekly during intervention phase; one month follow-up
  Therapeutic alliance/treatment acceptability. Higher scores indicate greater acceptability.
Treatment acceptability questions | one month follow-up
  Treatment acceptability. 6 questionnaire items on a Likert scale from strongly disagree to strongly agree. 4 open ended questions regarding treatment acceptability.
Items assessing parent knowledge of OCD, how to help their child, and confidence to help child | Weekly during baseline and intervention phase; one month follow up
  3 questionnaire items devised by study authors to assess parents' report of their knowledge and confidence to help their child to overcome OCD. Items scored from 0 (no new learning) to 5 (learned a lot)
Items assessing how much children have learned new information about their fears/ability to cope in feared situations | Weekly during intervention phase; one month follow up
  2 questionnaire items devised by study authors to assess parents' perceptions of whether their child had learned new information about their fears and their ability to cope in feared situations, without performing their compulsions. Items scored from 0 (no new learning) to 5 (learned a lot)

CONTACTS AND LOCATIONS:
Overall Officials: Kate N Harvey, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We are not able to make individual participant data available to other researchers.